CLINICAL TRIAL: NCT06435494
Title: C-PRO - The Effect of Cross-sectorial Use of Patient-Reported Outcomes for Patients With Chronic Degenerative Shoulder Conditions
Brief Title: Cross-sectorial Use of Patient-Reported Outcomes in Chronic Degenerative Shoulder Conditions
Acronym: C-PRO
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); VIVE - The Danish Center for Social Science Research (Other); The Novo Nordic Foundation (Other); Region Capital Denmark (Other); Mit Lægehus, Rødovre, Denmark (Unknown); Genoptræning og Rehabilitering, Rødovre Kommune, Denmark (Unknown); Center for Rehabilitering og Forebyggelse, Gentofte Kommune, Denmark (Unknown); Privathospitalet Danmark (Unknown)
Responsible Party: Principal Investigator, Anne Marie Nyholm, Principal investigator, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-23039139
Record Dates: First submitted 2024-05-16; First posted 2024-05-30 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Disease; Shoulder Impingement; Shoulder Osteoarthritis; Shoulder Frozen; Shoulder Capsulitis; Shoulder Bursitis; Shoulder Impingement Syndrome; Rotator Cuff Syndrome; Rotator Cuff Syndrome of Shoulder and Allied Disorders
MeSH Terms: conditions — Shoulder Impingement Syndrome; Bursitis

STUDY DESIGN:
Intervention Model Description: Patients evaluated and treated for a degenerative shoulder disorder will be randomised into two groups before first evaluation. For the intervention group, Patient reported outcomes (PRO) will be a part of the evaluation and follow-up of treatment. In the control group, it will not. Evaluation with PRO will be conducted every 3 months for 2 years follow-up.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to perform any blinding during collection and use of PRO data as part of the evaluation and treatment of the shoulder condition. However, following the end of PRO collection (and use), the following data collection and evaluation of the use of healthcare services and satisfaction with the treatment given will be performed with information of randomization blinded to the evaluators (VIVE).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): All patients will be asked to complete a number of questionaires: EQ5D-5L, a study specific questionaire (designed specifically for this study) and a shoulder-disease-specific questionaire (the Oxford Shoulder Score). For patients in the intervention group, the results of the questionaires will be accessable for patient and health-care professionals and will be used to illustrate the problems, make a prognostic model for the specific patient based on previous PRO results from other patients and will be used in monitoring the treatment of the patient.
  Interventions: Other: Systematic use of patient reported outcome measures in clinical work with the patients
- Control (No Intervention): All patients will be asked to complete a number of questionaires: EQ5D-5L, a study specific questionaire and a shoulder-disease-specific questionaire. For patients int he control group, this will be collected, but not accessed or used during the treatment of the patient. The data will be used in the final analyses of the study.

INTERVENTIONS:
Other: Systematic use of patient reported outcome measures in clinical work with the patients — Se description of the arms
  Arms: Intervention

SUMMARY:
This research project aims to test if systematic (extensive) use of patient-reported outcomes across treatment boundaries can

1. improve patients' and health professionals' understanding of individual patients' conditions and health changes,
2. improve indications for treatment,
3. strengthen patient empowerment, and
4. reduce patients' utilization of health services.

The study will be performed in the particular context of patients with chronic degenerative conditions of the shoulder. These patients are characterized by contact with numerous health professionals from different health sectors, such as general practitioner, physiotherapists and surgical referral centres, which challenges coherence and communication for the individual treatment decisions. The research project will be performed as a randomized controlled trial (RCT) with a 1-year inclusion period and two years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain with no acute trauma

Exclusion Criteria:

* Age <18 years
* Non-Danish citizenship
* Unable to understand written or spoken Danish
* Inability to master electronic means of communication and/or not having an electronic communication (E-boks)
* Employee at participating centre or other relation to participating health professionals that might affect independent consent
* Psychiatric conditions, mental conditions and substance abuse that might affect the ability to provide informed consent or responding to PROMs
* Disseminated malignant condition, other serious medical conditions or other life crisis where the focus on a shoulder research project is unreasonable
* Already included in the study with the contralateral shoulder

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment cost per change in life quality | From inclusion time and the 2 following years.
  The treatment cost during the study period expressed as the cost per improvement in life quality, similar to the cost per QALY (quality adjusted life years). The total cost will be calculated from hospital contacts, physiotherapy sessions and primary healthcare contacts. The EQ5D-5L will be used as a generic life quality measure. The primary outcome for the intervention and control group will be compared.

SECONDARY OUTCOMES:
Treatment cost per change in life quality stratisfied according to the specific shoulder diagnosis | From inclusion time and the 2 following years
  The same as primary outcome, but stratified according to the specific shoulder diagnosis
Patient satisfaction with the treatment of their shoulder problem | From inclusion time and the 2 following years
  Measured by questionaire (specifically the question "are you satisfied with the treatment fo your shoulder so far"?
Number of patients treated with surgery | From inclusion time and the 2 following years
  To evaluate if any difference in referral to surgery occurs between the intervention group and the control group, and analyse if any reasons for a difference can be identified
Number of contacts with either the hospital or the family doctor due to problems with the treated shoulder | From inclusion time and the 2 following years
  To evaluate if any difference in medical contacts due to the treated shoulder occurs between the intervention and the control groups, and analyse if any reasons for a difference can be identified
Number and types of complications during the treatment of the shoulder problem | From inclusion time and the 2 following years
  To evaluate if any difference in complications in relation to the treatment of the shoulder occurs between the intervention and the control groups, and analyse if any reasons for a difference can be identified
For patients still working: Number and duration (measured in days) of any periods of sick-leave/unemployment due to the shoulder problem | From inclusion time and the 2 following years
  To evaluate if any difference in employment-status and/or sick-leave occurs between the intervention and the control groups, and analyse if any reasons for a difference can be identified
Development in the PRO score, represented by Oxford Shoulder Score, over time for each specific shoulder disease | From inclusion time and the 2 following years
  To evaluate the development of PRO scores during a treatment of the included shoulder diseases with regards to the different treatment options, to create a reference for future treatments of these patients
PRO score, represented by Oxford Shoulder Score, as predictors? | From inclusion time and the 2 following years
  To evaluate if a PRO score can differentiate patients with regards to who might benefit from specific treatment regimens/effect of treatments measured by PRO
If use of systematic PRO scores, represented by Oxford Shoulder Score, changes the referral-pattern between the involved sectors | From inclusion time and the 2 following years
  To evaluate if PRO scores has the potential to be used to screen patients before making a referral between sectors
Health professionals' assessments of history and usefulness of the prognosis tools developed for this study (the Database setup in Procordo). | From inclusion time and the 2 following years
  To evaluate if the involved professionals experience any gain in the use of the PRO scores in the daily treatment of the patients. This will be evaluated at every visit with the patient by a questionaire to the treating professionals.
Patient satisfaction with the PRO score system build in the Database system (Procordo) | From inclusion time and the 2 following years
  Satisfaction and qualitative assessment of history and prognosis tool (intervention group only). This will be investigated by questionaire in relation to the completion of the PROs every 3 month during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Odgaard, MD, DrMed, Study Director — Rigshospitalet, Denmark; Anne M Nyholm, MD, PhD, Principal Investigator — University Hospital, Gentofte, Copenhagen; Bo S Olsen, MD, PhD, Study Chair — University Hospital, Gentofte, Copenhagen; Carsten B Juhl, PT, MPH, PhD, Study Chair — University Hospital, Gentofte, Copenhagen; Bente A Esbensen, Cand.cur., PhD, Study Chair — Rigshospitalet, Denmark
Locations (6):
- Denmark (6):
  - Department of Physiotherapy, Univesity Hospital Gentofte, Gentofte Municipality, Hellerup
  - Genoptræning og Rehabilitering, Rødovre Kommune, Rødovre Municipality, Rødovre
  - Privathospitalet Danmark, Charlottenlund
  - Department of rehabilitation, Gentofte Kommune, Hellerup
  - Division of shoulder and elbow surgery, Department of orthopaedics, Univesity Hospital Gentofte, Hellerup
  - Mit Lægehus, Rødovre Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nyholm AM, Esbensen BA, Westergaard CL, Kjellberg J, Juhl CB, Olsen BS, Odgaard A. Cross-sectoral use of Patient-Reported Outcomes (C-PRO)-the effect on the cost per improvement in quality of life for patients with chronic degenerative shoulder conditions-a protocol for a randomised controlled trial. Trials. 2025 Dec 12;27(1):47. doi: 10.1186/s13063-025-09329-0. PMID 41382298